CLINICAL TRIAL: NCT06318663
Title: Survivor Moms' Companion: A Perinatal PTSD Program
Brief Title: Survivor Mom Companion Comparison Study
Acronym: SMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ogechi Christine Kalu, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007685
Record Dates: First submitted 2024-03-11; First posted 2024-03-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Symptom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survivor Mom Companion Program (Active Comparator): Participants in the Survivor Moms' Companion intervention will complete a minimum of 4 Survivor Moms' Companion psychoeducational modules with weekly tutor support and will then complete an ending assessment. Sessions with tutors are conducted over the phone or in person at the Buffalo Prenatal and Perinatal Network and last for 45 minutes.
  Interventions: Other: Survivor Mom Companion
- Waitlist Control (Placebo Comparator): Participants in the waitlist control group will complete the baseline assessment over the phone, wait six weeks, and then complete the ending assessment. Those on the waitlist will then be offered the Survivor Moms' Companion intervention. Sessions with tutors are conducted over the phone or in person at the Buffalo Prenatal and Perinatal Network and last for 45 minutes.
  Interventions: Other: Survivor Mom Companion

INTERVENTIONS:
Other: Survivor Mom Companion — Weekly intervention sessions will follow the survivor Moms' Companion manualized modules. One module each week. The module centers on reinforcement of information introduced in each previous module, then emotional support, and referrals to additional services or specialists as needed. Participants in each session will practice applying knowledge and skills using the module's vignettes. Process guides prompt inquiry about in vivo management of post-traumatic stress disorder reactions and emotional and interpersonal responses to events since the last session. Each module may require 45 minutes of self-study before each session and 45 minutes of in-session time spent with the interventionist.

SUMMARY:
The overall goal of the SMC is to help reduce posttraumatic stress symptomology for pregnant persons with a history of trauma.

DETAILED DESCRIPTION:
The study is a pilot randomized waitlist-controlled trial that examines the preliminary efficacy of the SMC for reducing PTSD symptomology as compared to a waitlist control group. Also, it aims to assess the feasibility and acceptability of the SMC. It examines how changes in the theorized mechanisms (emotion regulation, interpersonal sensitivity) mediate the relationship between the intervention and PTSD symptomology.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* Currently pregnant or in the postpartum period
* Age 18 and older
* A history of trauma and PTSD
* Able to comprehend the study protocol and consent form and provide verbal consent and
* able to commit to a minimum of 4 weekly intervention sessions.

Exclusion Criteria:

* Non-English or non-Spanish-speaking,
* less than 18 years of age,
* those with psychotic conditions or developmental disabilities requiring guardianship,
* those with high-risk pregnancies necessitating extended bedrest or inpatient care, and
* those unable to commit to completing the intervention sessions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will self-identify.
Enrollment: 39 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Childhood Trauma Questionnaire | This will be administered prior to the intervention as part of the starting assessment.
  For eligibility screening we will use the 5 sentinel items from the Childhood Trauma Questionnaire. The higher the score is, the greater the severity of abuse for that scale. There are four categories of severity for each trauma type: None (minimal); Low (to Moderate); Moderate (to Severe); and Severe (to Extreme).
Primary Care Post Traumatic Stress Disorder Screen for Diagnostic and Statistical Manual of Mental Disorders-5 | This will be administered at the prior to the intervention as part of the starting assessment.
  The Primary Care post-traumatic stress Screen for Diagnostic and Statistical Manual of Mental Disorders is a 5-item screen designed to identify individuals with probable post-traumatic stress disorder. Primary Care Post Traumatic Stress Disorder considered "positive" if the respondent answers "yes" to any 3 items in the questions listed in the scale.
Adverse Childhood Experiences Questionnaire | This will be administered prior to the intervention as part of the starting assessment.
  Scale to assess the presence of childhood trauma. If the Adverse childhood experience score is 1-3 without Adverse Childhood Experience, the responder is at "intermediate risk" for toxic stress. If the Adverse childhood experience score is 1-3 and there is the likelihood of at least one Adverse childhood experience-associated condition, or if the Adverse childhood experiences score is 4 or higher, the responder is at "high risk" for toxic stress.
Post Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders | This will be administered prior to the intervention as part of the starting assessment and repeated after the intervention to assess any changes.
  Scale to assess presence of post-traumatic stress symptoms. Severity can be determined adding scores of each item together to determine a total score. A total score of 33 or higher may indicate severe post-traumatic stress disorder.
Dissociative Subtype of Post Traumatic Stress Scale | This will be administered prior to the intervention as part of the starting assessment and repeated after the intervention to assess any changes.
  Scale to assess dissociative symptoms. Each item on the measure is rated on a 5-point scale (0=Not at all; 1=Once or twice; 2=Almost every day; 3=About once a day, and 4=More than once a day). The total score can range from 0 to 32, with higher scores indicating greater severity of dissociative experiences.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | This will be administered prior to the intervention as part of the starting assessment and repeated after the intervention to assess any changes.
  A multipurpose instrument for screening and measuring severity of depression. In the scale 1-4 = minimal depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression and 20-27= severe depression. Thus, the higher the total score the higher the perceived level of depression.
State Trait Anger Expression Inventory | This will be administered prior to the intervention as part of the starting assessment and repeated after the intervention to assess any changes.
  A psychometric assessment that measures the experience and control of anger. scores are classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80). A higher score signifies higher anxiety.
Symptoms Checklist-90 Revised/Interpersonal Sensitivity Subscale | This will be administered prior to the intervention as part of the starting assessment and repeated after the intervention to assess any changes.
  Instrument help evaluate a broad range of psychological problem symptoms. Using a five-point scale ranging from "not at all" to "extremely", each item assesses the severity of distress the respondent experienced in the last 7 days. Each item is graded from 1 to 5 according to the severity (none, mild, moderate, severe and extreme). The scores of the items were regarded as extreme when the total is between 30-36.
Difficulties in Emotion Regulation Scale Short Form | This will be administered prior to the intervention as part of the starting assessment and repeated after the intervention to assess any changes.
  Covers four dimensions of emotional regulation; awareness and understanding of emotions, acceptance of emotions and the ability to engage in goal-directed behavior. All subscales are scored so that higher values reflect greater difficulty with emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mickey Sperlich, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Buffalo Prenatal-Perinatal Network, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Prins A, Bovin MJ, Smolenski DJ, Marx BP, Kimerling R, Jenkins-Guarnieri MA, Kaloupek DG, Schnurr PP, Kaiser AP, Leyva YE, Tiet QQ. The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5): Development and Evaluation Within a Veteran Primary Care Sample. J Gen Intern Med. 2016 Oct;31(10):1206-11. doi: 10.1007/s11606-016-3703-5. Epub 2016 May 11. PMID 27170304
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Wolf EJ, Mitchell KS, Sadeh N, Hein C, Fuhrman I, Pietrzak RH, Miller MW. The Dissociative Subtype of PTSD Scale: Initial Evaluation in a National Sample of Trauma-Exposed Veterans. Assessment. 2017 Jun;24(4):503-516. doi: 10.1177/1073191115615212. Epub 2015 Nov 23. PMID 26603115
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spielberger CD. Professional manual for the State-Trait Anger Expression Inventory-2 (STAXI-2). Odessa,FL: Psychological Assessment Resources; 1999.
- [Background] Derogatis LR, Lipman RS, Covi L. SCL-90. Administration, scoring and procedures manual-I for the R (revised) version and other instruments of the Psychopathology Rating Scales Series. Chicago: Johns Hopkins University School of Medicine; 1977.
- [Background] Kaufman EA, Xia M, Fosco G, Yaptangco M, Skidmore CR, Crowell SE. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and replication in adolescent and adult samples. Journal of Psychopathology and Behavioral Assessment. 2016 Sep;38(3):443-55. doi: 10.1007/s10862-015-9529-3
- [Background] Kelly PJ, Kyngdon F, Ingram I, Deane FP, Baker AL, Osborne BA. The Client Satisfaction Questionnaire-8: Psychometric properties in a cross-sectional survey of people attending residential substance abuse treatment. Drug Alcohol Rev. 2018 Jan;37(1):79-86. doi: 10.1111/dar.12522. Epub 2017 May 7. PMID 28480521

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT06318663/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT06318663/ICF_001.pdf